CLINICAL TRIAL: NCT05780528
Title: Mulligan Mobilization Versus Instrument Assissted Soft Tissue Mobilization In The Treatment Of Chronic Iateral Epicondylitis
Brief Title: Mulligan Mobilization Versus Instrument Assissted Soft Tissue Mobilization In Chronic Iateral Epicondylitis
Acronym: IASTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Yehia Helmy Abdelrahem, principle investigator nora yehia helmy Abdelrahem, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004235
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Lateral Epicondylitis
Keywords: instrumented assisted soft tissue mobilization; Mulligan Mobilization; lateral epiconylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: mulligan mobilization and instrumented-assisted soft tissue mobilization
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mulligan mobilization (Experimental): the patients will receive mulligan mobilization three times a week for four weeks
  Interventions: Other: mulligan mobilization; Other: conventional treatment
- instrumented assisted soft tissue mobilization (Experimental): the patients will receive instrumented assisted soft tissue mobilization three times a week for four weeks
  Interventions: Other: instrumented assisted soft tissue mobilization; Other: conventional treatment
- conventional treatment (Active Comparator): the patients will receive conventional treatment three times a week for four weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: mulligan mobilization — The patients will receive mobilization with movement technique of lateral glide. the patients will be in supine subject and pronate forearm, during the application of the lateral glide by the physiotherapist, each patient was asked to perform the closure of the fist (provocative but painless gesture in the execution of the technique) for 3 sets of 10 repetitions.
  Arms: mulligan mobilization
Other: instrumented assisted soft tissue mobilization — the participant will receive instrumented assisted soft tissue mobilization. The participant's elbow will rest on a table. A lubricant (Vaseline) will be applied to the skin around the elbow prior to treatment and the blade will be cleaned with an alcohol pad. First, the blade will be used to find the exact areas of restriction in the common extensor origin. Then the M2T blade will be used in the treatment planes 1, 2, and 3, to apply slow strokes along the muscle, without causing any discomfort or pain, from the muscle origin to its insertion (sweeping technique)
  Arms: instrumented assisted soft tissue mobilization
Other: conventional treatment — the patients will receive conventional treatment in the form of Ultrasound therapy, conventional transcutaneous electrical nerve stimulation (TENS) - hot pack - stretching and strengthening exercises and wrist rest splints

SUMMARY:
this study will be conducted to compare between mulligan mobilization and instrument assisted soft tissue mobilization on pain intensity, range of motion, hand grip strength, and hand function in the treatment of chronic lateral epicondylitis

DETAILED DESCRIPTION:
Lateral epicondylitis is one of the elbow conditions that affects about 1-3% of the population at large. It produces a heavy burden of workdays lost and residual impairments. Although many treatment modalities are used, few of them rest on scientific evidence and none has been proven more effective than the others. This lack of evidence on treatments for lateral epicondylitis may stem from several sources, including the possible self-limiting nature of the condition, the lack of pathophysiological data, the methodological shortcomings of available studies, and the existence of numerous factors influencing the outcome. The physiotherapeutic treatment has been shown to be effective. In general, it must include manual therapy to relieve the pain and improve the joint's range of motion (ROM), taking into account that it must be performed under the pain threshold. Mulligan mobilization with movement (MWM) is a modern technique developed by Mulligan for treating lateral epicondylitis (LE). Instrument-assisted soft tissue mobilization is a form of augmented soft tissue mobilization (IASTM) in which stainless steel instruments are utilized to apply controlled microtrauma to the affected soft tissues. sixty patients will be allocated randomly to three groups; the first one will receive mulligan mobilization with movement, the second one will receive instrument-assisted soft tissue mobilization and the third one will receive traditional therapy three times a week for four weeks

ELIGIBILITY:
Inclusion Criteria:

All patients will be diagnosed with chronic lateral epicondylitis from both genders.

Patients with chronic lateral epicondylitis were diagnosed by orthopedists. Positive clinical manifestation in all patients. Patients' age will be ranged from 18 to 80 years, Pain onset is more than 3 months. All participants must be medically stable and not be treated with analgesics or any medication which may cause misleading results.

All patients have a body mass index between 18.5 and 29.9 kg/m2.

Exclusion Criteria:

Patients who received an intra-articular injection for a duration of less than 3 months.

Patients receiving oral or injected corticosteroids for the last 3 months at least.

History of elbow surgery/fracture. Acute synovitis/arthritis including infectious. Presence of malignancy. Pregnancy. Patients with, topical lesions, contact dermatitis, and a history of cutaneous hypersensitivity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-25 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  pain will be measured by visual analogue scale. It is a vertical or horizontal 100 mm line graduated by different levels of pain, starting from 0 (no pain) till 100 (worst pain)
shoulder disability | up to four weeks
  The Arabic version of Disabilities of arm, shoulder, and hand (DASH) will be used for assessing shoulder function.DASH questionnaire includes 11 items with score from 0 to 100. A score of 0 represents no disability, while a score of 100 represents the most sever

SECONDARY OUTCOMES:
range of motion | up to four weeks
  elbow and wrist range of motion will be measured by universal goniometer
hand grip strength | up to four weeks
  Hand held dynamometer will be used to measure hand grip strength